CLINICAL TRIAL: NCT07398898
Title: Use of New Technologies in Dentistry
Brief Title: Use of Augmented Reality Glasses and Noise-Cancelling Headphones to Reduce Dental Anxiety in Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KB/98/2023
Record Dates: First submitted 2025-05-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety; Music Therapy; Oral Surgical Procedures
Keywords: dental anxiety; Music therapy; augmented reality; active noise cancelling; maxillofacial surgery; Dental phobia; audiovisual distraction; dental fear; perioperative anxiety; STAI; galvanic skin response; relaxation techniques

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: a control group (no audiovisual intervention), an intervention group using noise-cancelling headphones playing relaxing music, or an intervention group using augmented reality (AR) glasses displaying relaxing video with the same music. Each participant receives only one intervention throughout the dental procedure. No crossover between groups will occur.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants, regardless of group assignment, will undergo the same physiological monitoring using a wrist-worn device that records skin conductance and heart rate via adhesive electrodes placed on the hand. This standardized setup enhances participant masking by making the procedure appear uniform across all groups. In addition, participants in the control group will receive sensory placebo devices-either non-functioning headphones or non-digital protective glasses-designed to resemble the active interventions. Outcomes will be assessed by blinded data analysts. Care providers and investigators will not be blinded due to the visible nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AR Glasses with Video and Music (Experimental): Participants in this group will wear lightweight augmented reality (AR) glasses during the dental procedure. The glasses display calming, nature-themed visual content accompanied by relaxing instrumental music. The audiovisual material is presented continuously throughout the procedure. The goal of this intervention is to provide immersive distraction to reduce dental anxiety and physiological stress. Physiological signals (such as skin conductance and heart rate) will be recorded simultaneously using wearable sensors. The audiovisual setup is noninvasive, requires no interaction from the patient, and allows real-time communication with the dental team.
  Interventions: Device: AR Glasses with Video and Music
- ANC Headphones with Music (Experimental): Participants in this group will wear over-ear active noise-cancelling headphones during the dental procedure. The headphones continuously play relaxing instrumental music, and their active noise cancellation (ANC) function helps mask clinical sounds such as drilling or suction. The intervention aims to reduce dental anxiety and enhance patient comfort by limiting auditory stressors. Physiological signals (including skin conductance and heart rate) will be recorded using wearable sensors throughout the procedure. The music does not interfere with communication, and the device can be adjusted to allow interaction with the clinical staff.
  Interventions: Device: ANC Headphones with Music
- Control Group with Sensory Placebo (Placebo Comparator): Participants in the control group will receive one of two types of sensory placebo during the dental procedure: (1) non-functional over-ear headphones that do not play music or provide noise cancellation, or (2) protective glasses resembling AR glasses that do not display any image or produce sound. All participants will wear the same physiological sensors on the wrist and hand, regardless of group. The purpose of this design is to maintain procedural uniformity and partially mask group assignment. No audiovisual stimulation is provided in this group.
  Interventions: Device: Sensory Placebo Devices

INTERVENTIONS:
Device: AR Glasses with Video and Music — Participants wear augmented reality (AR) glasses that display calming nature-themed video content accompanied by relaxing music. The audiovisual content is presented throughout the dental procedure. The glasses are non-obstructive and allow patient-dentist communication. The purpose is to provide immersive distraction to reduce anxiety and physiological stress.
  Other Names: Augmented reality audiovisual distraction
  Arms: AR Glasses with Video and Music
Device: ANC Headphones with Music — Participants wear over-ear noise-cancelling headphones during the dental procedure. The headphones continuously play relaxing music and reduce environmental dental noise via active noise cancellation (ANC). The goal is to reduce anxiety and improve patient comfort during treatment.
  Other Names: Active Noise Cancelling Headphones audio distraction
  Arms: ANC Headphones with Music
Device: Sensory Placebo Devices — Participants in the control group receive a sensory placebo: either protective glasses that resemble AR glasses but do not display video, or over-ear headphones that do not emit sound or noise cancellation. This simulates the intervention experience without actual audiovisual input and helps partially blind participants to their group assignment.
  Other Names: Placebo Glasses or Headphones
  Arms: Control Group with Sensory Placebo

SUMMARY:
This study investigates whether new audiovisual technologies can help reduce anxiety and stress experienced by adult patients during dental procedures. Dental fear and anxiety are common barriers to receiving proper oral care. This randomized controlled trial aims to explore whether the use of specific devices-augmented reality (AR) glasses and noise-cancelling (ANC) headphones-can improve patient comfort and decrease physiological signs of stress during dental treatment.

Participants in this study will undergo a standard dental procedure. In addition, they will be randomly assigned to one of three groups: a control group (no audiovisual intervention), a group using ANC headphones that play relaxing music during the procedure, or a group using AR glasses that display relaxing visual scenes along with the same music.

Before the procedure, each participant will complete a psychological questionnaire (STAI) to assess their level of anxiety. During the procedure, physiological stress will be monitored using sensors that track parameters such as skin conductance (GSR) and heart rate. After the treatment, patients will be asked to rate their pain level and describe their experience with or without the audiovisual intervention.

The goal is to better understand the effectiveness of non-pharmacological methods in reducing anxiety and stress in adult dental patients. Participation in the study is entirely voluntary and will not affect the quality or availability of dental care. Patients may withdraw at any time without consequences. The study also collects basic demographic information and patient feedback to evaluate potential factors that may influence anxiety levels.

By testing new immersive tools such as AR glasses and ANC headphones in a real clinical setting, this research may contribute to improving patient well-being and enhancing the dental care experience.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the effectiveness of two audiovisual interventions-augmented reality (AR) glasses with immersive video and relaxing music, and over-ear headphones with active noise cancellation (ANC) and relaxing music-for reducing anxiety and improving the overall patient experience during dental surgical procedures.

Dental anxiety is a major barrier to effective oral healthcare and is associated with increased stress, physiological arousal, and patient avoidance behaviors. This trial is designed to test whether immersive audiovisual distraction can significantly lower anxiety and stress levels, as measured both subjectively (via standardized questionnaires) and objectively (via physiological metrics such as skin conductance and heart rate).

A total of up to 250 adult patients will be enrolled, with a planned final analysis sample of 192 participants equally divided into three arms: (1) AR glasses with immersive nature video and relaxing music (VITURE Pro XR); (2) over-ear headphones with ANC (Apple AirPods Max) playing relaxing music; and (3) a control group using non-functional sensory placebo (protective glasses or non-playing headphones) but receiving identical physiological monitoring. All patients undergo routine dental procedures, mostly surgical (e.g., extractions, curettage), as scheduled at the University Dental Center of the Medical University of Warsaw (WUM).

Randomization will be computer-generated using simple randomization (1:1:1) via a pre-generated allocation list in Microsoft Excel. Random assignment will occur prior to the procedure by the lead researcher who is otherwise blinded to the data collection. Participants will not be told which intervention is expected to be most effective.

All participants are fitted with a wrist-worn physiological sensor (Shimmer3 GSR+) with palm electrodes and an optical pulse probe on the fingertip. These devices continuously monitor skin conductance and pulse rate during the entire dental procedure. Measurements are recorded digitally using ConsensysPRO software and stored in anonymized CSV format on a secure, dedicated study computer. No personally identifiable information is stored in analysis files.

Primary outcome is the change in subjective anxiety as measured by the STAI-Y1 questionnaire, administered before and after the dental procedure. Secondary outcomes include skin conductance level (GSR), heart rate (HR), post-procedure pain intensity (VAS), and qualitative feedback on intervention experience. Sociodemographic data (age, sex, education level, prior dental experiences) will be collected at baseline. The duration of the procedure, equipment status, and patient behavior are also documented in observation notes.

Quality assurance will include cross-verification of physiological data against time-stamped observation logs. Any anomalies (e.g., loss of signal due to electrode detachment or excessive motion artifacts) will be documented, and those cases flagged for potential exclusion in per-protocol analysis. All enrolled participants will be included in intention-to-treat analysis unless withdrawn or consent is revoked.

Randomization, participant enrollment, and intervention delivery are overseen by the study director (doctoral candidate) and supervised by the principal investigator affiliated with the Department of Oral Mucosal and Periodontal Diseases, WUM. The protocol has been approved by the institutional bioethics committee (reference: KB/98/2023). Minimal risk is anticipated, as interventions are non-invasive, optional, and reversible. Participants are informed that refusal to participate will not affect their treatment in any way.

Data will be handled in compliance with GDPR and institutional regulations. Cases with missing data or interrupted recordings will be documented with reason codes. Visual and auditory materials used in the intervention have been vetted for calmness and neutrality to avoid emotional triggers. Participants may withdraw at any time.

This study seeks to identify scalable, evidence-based strategies to mitigate dental anxiety using modern, patient-friendly technologies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Qualified for one of the following dental procedures: supragingival scaling, curettage, tooth extraction, or caries cavity preparation and restoration
* Provided written informed consent
* Agreed to random allocation to one of the study groups
* Able to understand and complete the STAI questionnaire and VAS pain scale

Exclusion Criteria:

* Acute dental pain at the time of the procedure
* Teeth qualified for resection
* Pregnancy
* Diagnosis of cerebral palsy
* Epilepsy with seizures in the past 6 months
* Use of hearing aids
* Severe vision impairment
* Non-cooperative behavior or inability to understand the study questionnaires
* Absence on the scheduled procedure date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Anxiety Level (STAI Score) | Immediately after the dental procedure
  Change in subjective anxiety assessed using the State-Trait Anxiety Inventory (STAI), Form Y-1. Participants complete the questionnaire immediately before (baseline) and immediately after the dental procedure. The outcome is defined as the difference between post- and pre-procedure STAI-Y1 scores. Scores range from 20 to 80, with higher scores indicating greater anxiety. The difference in pre- and post-procedure scores will be calculated and compared across study arms.

SECONDARY OUTCOMES:
Skin Conductance Level (GSR) During Dental Procedure | Perioperative (during dental procedure)
  Measurement of skin conductance level (GSR), reflecting autonomic nervous system activity and physiological stress response. Conductance in microsiemens (μS) is recorded continuously using a wrist-worn sensor with electrodes adhered to the palm. Average GSR values over the treatment period will be compared between study arms.
Heart Rate Monitoring During Dental Procedure | Perioperative (during dental procedure)
  Continuous non-invasive measurement of heart rate using a fingertip optical pulse sensor (based on photoplethysmography). The sensor tracks real-time pulse rate, reflecting cardiovascular response to stress. Mean heart rate across the procedure duration will be analyzed between groups.
Self-Reported Pain During Procedure (VAS Score) | Immediately after the dental procedure
  Subjective pain intensity will be measured using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst imaginable pain). Participants will rate their perceived pain immediately after the procedure. Scores will be compared between arms.

OTHER OUTCOMES:
Participant Feedback on Audiovisual Setup (Exploratory) | Immediately after the dental procedure
  An optional open-ended field will collect spontaneous patient feedback regarding audiovisual or placebo devices. Responses will not be scored quantitatively but may be used for exploratory qualitative assessment of user experience and perceived comfort. No numerical rating scale is used for this measure.
Exploratory Analysis of Sociodemographic Characteristics | Once, at enrollment
  Data on sex, age, education level, prior negative dental experiences, and time since last dental visit will be collected. These characteristics will be used to explore potential moderators of treatment effect. No formal hypothesis is defined.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kowalski, Associate Professor, MD, PhD, Principal Investigator — Medical University of Warsaw; Jakub Bereziewicz, MSc, Study Director — Medical University of Warsaw
Locations (1):
- University Dental Center, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) is currently undecided. IPD sharing may depend on institutional policies of the Medical University of Warsaw, ethical approval, and data protection considerations. At this stage, no repository or mechanism for de-identified data sharing has been established.

REFERENCES:
- See also: Related Info — https://stomatologia.wum.edu.pl/

DOCUMENTS (1):
  • Informed Consent Form (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT07398898/ICF_000.pdf